CLINICAL TRIAL: NCT02734901
Title: Effects of Acute Red Raspberry Consumption on Vascular Function in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Rapsberry; 15-038 (Other: CTSU)
Record Dates: First submitted 2016-03-09; First posted 2016-04-12 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: polyphenols; vascular function; endothelial function; raspberry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 400 g frozen raspberries (Active Comparator): Red raspberry beverage Acute intake of 600 mL (1x daily)
  Interventions: Dietary Supplement: 400 g frozen raspberries
- 200 g frozen raspberries (Active Comparator): Red raspberry beverage Acute intake of 600 mL (1x daily)
  Interventions: Dietary Supplement: 200 g frozen raspberries
- Placebo control (Placebo Comparator): Raspberry deprived supplement Acute intake of 600 mL (1x daily)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 400 g frozen raspberries — 1x daily intake of 600 mL red raspberry beverage
  Arms: 400 g frozen raspberries
Dietary Supplement: 200 g frozen raspberries — 1x daily intake of 600 mL red raspberry beverage
  Arms: 200 g frozen raspberries
Dietary Supplement: Placebo — 1x daily intake of 600 mL raspberry deprived supplement
  Arms: Placebo control

SUMMARY:
Accumulating evidence from epidemiological and human intervention studies indicates that the cardiovascular health benefits of diets rich in fruits and vegetables are (in part) related to their (poly)phenol content. Raspberries are rich in phenolic and polyphenolic compounds, in particular procyanidins, ellagitannins and anthocyanins, but also phenolic acids. At present, a small number of randomized controlled trials investigating the effects of berry (poly)phenols on validated surrogate markers of cardiovascular disease risk have shown promising results. However, to date, very few human studies have specifically investigated the effects of raspberry (poly)phenols on cardiovascular function in healthy subjects. Moreover, ellagitannin-derived metabolites are believed to persist for a long period of time in the blood and urine. Therefore, the investigators will investigate the presence of plasma and urinary raspberry-derived metabolites 24h post-consumption. To the investigators knowledge, the effects of red raspberry consumption on vascular function in humans have not been investigated before. This information is necessary for the planning of long-term studies aiming to assess the potential beneficial effects of raspberries,. Therefore, this study aims to investigate the potential role of red raspberry (poly)phenols in the modulation of vascular function by monitoring changes in vascular function together with the major (poly)phenol derivatives/metabolites in plasma.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects (no clinical signs or symptoms of cardiovascular disease)

Exclusion Criteria:

* Cardiovascular disease
* acute inflammation
* cardiac arrhythmia
* renal failure
* heart failure (NYHA II-IV)
* diabetes mellitus
* C - reactive protein > 05 mg/dL
* malignant disease
* raspberry allergy/intolerance
* hypotension (≤100 / 60 mm Hg)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 2 hour and 24 hour in Endothelial function | Baseline, 2 hour and 24 hour
  measured by flow mediated dilation (FMD) on baseline at 2 and 24 hour postconsumption

SECONDARY OUTCOMES:
Change from baseline to 2 hour and 24 hour in Pulse wave velocity | Baseline, 2 hour and 24 hour
  measured by sphygmomanometer SphygmoCor on baseline at 2 and 24 hours postconsumption
Change from baseline to 2 hour and 24 hour in Central blood pressure | Baseline, 2 hour and 24 hour
  measured by sphygmomanometer SphygmoCor on baseline at 2 and 24 hours postconsumption
Peripheral blood pressure | Baseline, 2 h and 24 h
  measured by automatic sphygmomanometer on baseline at 2 and 24 hours postconsumption
Change from baseline to 2 hour and 24 hour in Heart rate | Baseline, 2 hour and 24 hour
  measured by SphygmoCor on baseline at 2 and 24 hours postconsumption

OTHER OUTCOMES:
Change from baseline to 2 hour and 24 hour in Polyphenol metabolites in blood plasma | Baseline, 2 hour and 24 hour
  measured by ultra-performance liquid chromatography/quadrupole-time-of-flight mass-spectrometry (UPLC-Q-TOF MS ) on baseline at 2 and 24 hours postconsumption
Change from baseline to 2 hour and 24 hour in Polyphenol metabolites in urine | Baseline, 2 hour and 24 hour
  measured by ultra-performance liquid chromatography/quadrupole-time-of-flight mass-spectrometry (UPLC-Q-TOF MS ) on baseline at 2 and 24 hours postconsumption

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf; Christian Heiss, MD, Principal Investigator — Division of Cardiology, Pulmonology and Vascular Medicine, University Hospital Duesseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, University Hospital Duesseldorf, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Istas G, Feliciano RP, Weber T, Garcia-Villalba R, Tomas-Barberan F, Heiss C, Rodriguez-Mateos A. Plasma urolithin metabolites correlate with improvements in endothelial function after red raspberry consumption: A double-blind randomized controlled trial. Arch Biochem Biophys. 2018 Aug 1;651:43-51. doi: 10.1016/j.abb.2018.05.016. Epub 2018 May 24. PMID 29802820